CLINICAL TRIAL: NCT01454206
Title: Integration of Internet-facilitated Screening, Brief Intervention, Referral to Treatment (iSBIRT) for Teen Drug Use Into a Pediatric Network
Brief Title: Integration of (iSBIRT) for Teen Drug Use Into a Pediatric Network
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The project was not funded
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CeASAR app RFADA12008
Record Dates: First submitted 2011-10-05; First posted 2011-10-18 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Substance Use
Keywords: cannabis abuse; alcohol abuse; substance abuse
MeSH Terms: conditions — Substance-Related Disorders; Marijuana Abuse; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (No Intervention)
- iSBIRT (Experimental): Participants will receive the internet-facilitated screening, brief intervention and referral to treatment (iSBIRT intervention)
  Interventions: Behavioral: iSBIRT

INTERVENTIONS:
Behavioral: iSBIRT — Participants will be screened for substance use, view information about the health effects of substance use on the computer, and receive advice from the primary care provider regarding the health effects of substance use. Those found to be at "high risk" will complete an internet-based program encouraging them to change their substance use.
  Arms: iSBIRT

SUMMARY:
The Goal of this project is to integrate a previously-tested internet-facilitated Screening, Brief Intervention, and Referral to Treatment (iSBIRT) system for adolescent substance use into a large network of primary care offices, the Pediatric Practices of Children's Hospital Boston (PPOC).

ELIGIBILITY:
Inclusion Criteria:

* 12-18 year olds
* Coming for non-emergent care
* Access to a private computer
* Have email address

Exclusion Criteria:

* Not available for follow-up questionnaires
* Unable to read or understand English at a 6th grade reading level
* Medically or emotionally unstable on the day of the visit

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Provider attitude toward iSBIRT | 12 months post baseline
  We will evaluate providers' acceptance of and attitude toward integrating iSBIRT into their practices.

SECONDARY OUTCOMES:
Youth connectedness to provider | Baseline
  We will measure adolescents' attitudes toward their providers' advice regarding the health effects of substance use given during the visit
iSBIRT sustainability | 12 months post
  We will measure rates of continued use of iSBIRT by practices 12 months after iSBIRT recruitment and implementation ends
Change in rates of adolescent substance use | 3 months post baseline
  We will measure the change in rates of adolescent substance use from baseline to 3 months post study visit.
Change in rates of adolescent substance use | 6 months post baseline
  We will measure the change in rates of adolescent substance use from baseline to 6 months post study visit.
Change in rates of adolescent substance use | 12 months post baseline
  We will measure the change in rates of adolescent substance use from baseline to 12 months post study visit.

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- See also: Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org